CLINICAL TRIAL: NCT04488094
Title: A Phase 2, Open-label, Non-randomized, Single Center Study to Explore Diagnostic Performance of [18F]FSPG PET/CT for the Assessment of Acute Allograft Rejection After Heart or Liver Transplantation
Brief Title: Diagnostic Validity of [18F]FSPG PET for the Assessment of Acute Rejection After Heart or Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae Hyuk Moon, Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FSPG-1902
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Graft Rejection; Heart Transplantation; Liver Transplantation
Keywords: Graft Rejection; Heart Transplantation; Liver Transplantation; Positron-Emission Tomography; Diagnostic Imaging
MeSH Terms: interventions — 4-(3-fluoropropyl)glutamic acid

STUDY DESIGN:
Intervention Model Description: Patients suspected of having acute allograft rejection after heart transplantation (HT, n = 10) or liver transplantation (LT, n = 10)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart transplantation (Experimental): Patients suspected of having acute heart allograft rejection after heart transplantation will receive a single IV injection of [18F]FSPG
  Interventions: Drug: [18F]FSPG
- Liver transplantation (Experimental): Patients suspected of having acute liver allograft rejection after heart transplantation will receive a single IV injection of [18F]FSPG
  Interventions: Drug: [18F]FSPG

INTERVENTIONS:
Drug: [18F]FSPG — A radioactive dose of 200 MBq of the study drug with a total quantity of ≤ 100 µg will be administered as slow intravenous bolus injection over up to 60 seconds. PET/CT examinations will be performed at 60-75 min after the administration of [18F]FSPG.
  Other Names: FSPG

SUMMARY:
The a series of clinical studies of [18F]FSPG PET/CT showed that [18F]FSPG is safe and promising PET tracer for detecting inflammation with favorable biodistribution and pharmacokinetics in patients. By using [18F]FSPG, which targets system xCˉ, a key player in the active phase of inflammation, the goal of this phase 2 study is to evaluate diagnostic validity of [18F]FSPG PET/CT to detect allograft rejection after heart and liver allograft, where conventional imaging has limitations. Diagnostic efficacy of [18F]FSPG PET/CT will be determined in comparison with histologic evaluation of allograft biopsy. Other critical questions including whether quantitative measures of [18F]FSPG uptake is associated with the severity of rejection, inter-reader variability of [18F]FSPG PET/CT, and safety assessment will be also evaluated.

DETAILED DESCRIPTION:
This open label, non-randomized, single center, single-dose exploratory study is designed to obtain imaging assessments using PET/CT with [18F]FSPG in patients with heart transplantation (HT, n = 10) and liver transplantation (LT, n = 10). Subjects who underwent or scheduled to undergo biopsy for histologic diagnosis of acute rejection will be enrolled.

The study comprises 3 periods: screening, treatment, and follow-up. The screening period starts with the subject's signature on the informed consent form and ends with assignment to treatment that is inclusion of the subject for treatment. The treatment period starts with baseline measurements, and ends with the last measurement/procedure on the day following injection of 200 MBq of [18F]FSPG. The follow-up period contains the end-of-study interview. Key measurement is the PET/CT image acquisition about one hour after the single injection of [18F]FSPG. For evaluation of safety, adverse events (AE) will be monitored and recorded during the study period.

This study will be monitored regularly by a clinical research associate from the sponsor or a designated contract research organization. Data quality and study integrity will be assessed. The investigator will document the items that are required to evaluate the study in the subject files. Data required according to this protocol are to be recorded on the case report forms provided by the sponsor as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged between 19 and 79 years and male or female of any race/ethnicity.
* Subject received heart transplantation or liver transplantation at least 30 days prior to screening
* Subject underwent or is scheduled to undergo biopsy for histologic diagnosis of acute rejection within 7 days prior to or after the planned [18F]FSPG PET/CT administration.

Exclusion Criteria:

* Subject or subject's legally acceptable representative does not provide written informed consent.
* Dose escalation of the current immunosuppressant drugs or starting a new immunosuppressant is scheduled from the study enrollment to the scheduled day of biopsy, or 24 hours after [18F]FSPG administration
* Female subject is pregnant or nursing. Exclusion of the possibility of pregnancy is made by one of the following: 1) Woman is physiologically post-menopausal (cessation of menses for more than 2 years), 2) woman is surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy, or 3) if the woman is of childbearing potential, a serum or urine pregnancy test performed within 24 hours immediately prior to administration of [18F]FSPG has to be negative and the women is advised to apply contraceptive measures during her participation in this study.
* Subject has concurrent severe and/or uncontrolled and/or unstable medical disease (e.g. congestive heart failure, acute myocardial infarction, severe pulmonary disease, chronic renal or hepatic disease which could compromise participation in the study) in the judgment of the investigator.
* Subject is a relative of the investigator, student of the investigator or otherwise dependent.
* Subject has received any investigational drugs or devices within four weeks prior to the study enrollment or within 24 hours after administration of [18F]FSPG.
* Subject has been previously included in this study.
* Subject has any other condition or personal circumstances that, in the judgment of the investigator, might make collection of complete data difficult or impossible.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of qualitative [18F]FSPG PET/CT interpretation for the diagnosis of patients with histologic evidence of acute allograft rejection | within 7 days of [18F]FSPG PET/CT
  sensitivity = (the number of [18F]FSPG PET/CT-positive patients divided by the number of rejection positive patients on the histological evaluation) x 100; specificity = (the number of [18F]FSPG PET/CT-negative patients divided by the number of rejection negative patients on the histological evaluation) x 100

SECONDARY OUTCOMES:
Association between quantitative [18F]FSPG uptake and histologic grade of rejection | within 7 days of [18F]FSPG PET/CT
  The association between [18F]FSPG uptake and the histologic grades of rejection activity using Pearson or Spearman rank correlation coefficient
Inter-reader variability | within 1 day of [18F]FSPG PET/CT
  Inter-reader variability of [18F]FSPG uptake score measured using the kappa statistic
Incidence of treatment emergent adverse events | From the administration of [18F]FSPG to one day after [18F]FSPG PET/CT
  Number of participants with treatment emergent adverse events graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0)
Blood pressure | Pre-treatment and three hours after the administration of [18F]FSPG
  mmHg
Heart rate | Pre-treatment and three hours after the administration of [18F]FSPG
  beats/minute
Body temperature | Pre-treatment and three hours after the administration of [18F]FSPG
  Celsius
Physical examination | Pre-treatment and three hours after the administration of [18F]FSPG
  The limited physical examination will comprise: general appearance, skin, neck, lungs, heart, abdomen, and a limited neurological examination (mental status, motor strength and sensor perception)
Blood tests for safety | Pre-treatment and three hours after the administration of [18F]FSPG
  The clinical laboratory safety parameters to be assessed are as follows: glutamate pyruvate transaminase (GPT/ALAT), glutamate-oxaloacetate transaminase (GOT/ASAT), alkaline phosphatase, total bilirubin, creatinine, potassium, sodium, total protein, blood urea nitrogen (BUN), albumin

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyuk Moon, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koglin N, Mueller A, Berndt M, Schmitt-Willich H, Toschi L, Stephens AW, Gekeler V, Friebe M, Dinkelborg LM. Specific PET imaging of xC- transporter activity using a (1)(8)F-labeled glutamate derivative reveals a dominant pathway in tumor metabolism. Clin Cancer Res. 2011 Sep 15;17(18):6000-11. doi: 10.1158/1078-0432.CCR-11-0687. Epub 2011 Jul 12. PMID 21750203
- [Background] Chae SY, Choi CM, Shim TS, Park Y, Park CS, Lee HS, Lee SJ, Oh SJ, Kim SY, Baek S, Koglin N, Stephens AW, Dinkelborg LM, Moon DH. Exploratory Clinical Investigation of (4S)-4-(3-18F-Fluoropropyl)-L-Glutamate PET of Inflammatory and Infectious Lesions. J Nucl Med. 2016 Jan;57(1):67-9. doi: 10.2967/jnumed.115.164020. Epub 2015 Oct 15. PMID 26471694
- [Background] Baek S, Choi CM, Ahn SH, Lee JW, Gong G, Ryu JS, Oh SJ, Bacher-Stier C, Fels L, Koglin N, Hultsch C, Schatz CA, Dinkelborg LM, Mittra ES, Gambhir SS, Moon DH. Exploratory clinical trial of (4S)-4-(3-[18F]fluoropropyl)-L-glutamate for imaging xC- transporter using positron emission tomography in patients with non-small cell lung or breast cancer. Clin Cancer Res. 2012 Oct 1;18(19):5427-37. doi: 10.1158/1078-0432.CCR-12-0214. Epub 2012 Aug 14. PMID 22893629
- [Background] Baek S, Mueller A, Lim YS, Lee HC, Lee YJ, Gong G, Kim JS, Ryu JS, Oh SJ, Lee SJ, Bacher-Stier C, Fels L, Koglin N, Schatz CA, Dinkelborg LM, Moon DH. (4S)-4-(3-18F-fluoropropyl)-L-glutamate for imaging of xC transporter activity in hepatocellular carcinoma using PET: preclinical and exploratory clinical studies. J Nucl Med. 2013 Jan;54(1):117-23. doi: 10.2967/jnumed.112.108704. Epub 2012 Dec 11. PMID 23232273